CLINICAL TRIAL: NCT04488497
Title: Optimization of Hyperlipidemia Management Among Patients With Rheumatoid Arthritis: A Patient-centered Intervention Development
Brief Title: Cardiovascular Risk Assessment for Patients With Rheumatoid Arthritis Arthritis:
Acronym: CARE RA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: 1703018030; K23AR068449 (NIH)
Record Dates: First submitted 2020-07-22; First posted 2020-07-28 (Actual); Results first posted 2025-10-24 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-10

CONDITIONS: Rheumatoid Arthritis; Cardiovascular Diseases; Hyperlipidemias
Keywords: Self-efficacy; Patient activation; Social Cognitive Theory; Peer coaches
MeSH Terms: conditions — Arthritis, Rheumatoid; Cardiovascular Diseases; Hyperlipidemias; Patient Participation | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Peer coach guided online learning program (Experimental)
  Interventions: Behavioral: Cardiovascular Risk Assessment for Patients with Rheumatoid Arthritis
- Self-administered online learning program (Active Comparator)
  Interventions: Behavioral: Standard of care

INTERVENTIONS:
Behavioral: Cardiovascular Risk Assessment for Patients with Rheumatoid Arthritis — This intervention will help people with RA get tested for hyperlipidemia so that they can later discuss with their physician how to better treat their increased risk for cardiovascular disease.
  Arms: Peer coach guided online learning program
Behavioral: Standard of care — Participants in this group will not receive peer coaches calls. They will receive additional educational materials about CVD risk and the regular care provided by their doctors.
  Arms: Self-administered online learning program

SUMMARY:
One of the greatest success stories in rheumatology - the achievement of rheumatoid arthritis (RA) remission - is tempered by the fact that individuals with RA are dramatically under evaluated and under treated to reduce the risk for heart attacks and strokes. This project will build the foundation for an intervention that will test the hypothesis that the patient-centered intervention tailored to patients with RA to improve hyperlipidemia screening and treatment, thereby decreasing the risk for heart attacks and strokes.

The aims of this proposal are:

Aim 1: To identify patient and physician barriers to lower the risk for heart attacks and strokes in patients with RA.

Aim 2: To develop an intervention designed to optimize lipid screening and management in RA patients. This will consist of patient education and a decision support program to facilitate screening for hyperlipidemia (high cholesterol level) or initiation of medications to lower cholesterol (primary outcome) and self-efficacy (level of confidence in performing a task) in taking medications to lower cholesterol secondary outcome).

Aim 3: To pilot test the efficacy and feasibility of intervention developed in Aim 2. The investigators will apply methods related to clinical trials to test the feasibility of the newly developed intervention.

ELIGIBILITY:
Inclusion Criteria:

* Have RA
* Age between 40 and 75 years (inclusive)
* Provide a date of their next appointment with their rheumatologist or other physician on their care team
* Willing to work with a peer coach
* Speaks English
* Have a phone
* Has access to the internet
* Resides or lives in the US

Exclusion Criteria:

* Do not have rheumatoid arthritis
* Younger than age 40 or older than age 75
* Taking a statin
* No known history of diabetes
* No known history of CVD defined by:

  * Open heart surgery
  * Coronary angioplasty
  * History of heart failure
  * History of heart attack or stroke

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2021-01-27 (Actual); Primary Completion 2024-11-06 (Actual); Study Completion 2024-11-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Iris Navarro-Milan, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Weiner J, Lui G, Brown M, Paez YD, Fritz S, Sydnor-Campbell T, Allen A Jr, Jabri A, Venkatachalam S, Gavigan K, Nowell WB, Curtis JR, Fraenkel L, Safford M, Navarro-Millan I. Protocol for the pilot randomized trial of the CArdiovascular Risk assEssment for Rheumatoid Arthritis (CARE RA) intervention: a peer coach behavioral intervention. Pilot Feasibility Stud. 2022 Apr 15;8(1):84. doi: 10.1186/s40814-022-01041-z. PMID 35428359

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period was from January 2021 to October 2024. Recruitment was facilitated via registries provided by the partnering organizations ArthritisPower, BuildClinical, and the BendCare Patient Network. The EHR Data and Reporting system TRAC was used to generate patient lists of potentially eligible patients from partnering surgeons.
  The first participant was enrolled on January 27, 2021 and the last participant was enrolled on June 5th, 2024.
Groups:
- Peer Coach Guided Online Learning Program: The CARE RA intervention consists of 3 components: peer support, patient activation, and online education via the patient activation learning website (PALS). Over the course of 5 weeks before their upcoming physician's appointment, participants met with a peer coach (a person with RA who has been trained on delivering the content of the CARE RA intervention to another person with RA) for weekly 30-45 minute one-on-one telephonic sessions to reinforce key points in the CARE RA curriculum within the PALS.
- Self-administered Online Learning Program (Control): The self-administered control arm consists of a tutorial on how to use the Patient Activated Learning System (PALS) followed by self-driven completion of the CARE RA curriculum within the PALS over the course of 5 weeks before their upcoming physician's appointment.
Period: Randomization/Baseline Assessment
Arm/Group | Peer Coach Guided Online Learning Program | Self-administered Online Learning Program (Control)
Started | 49 | 52
Completed | 47 | 49
Not Completed | 2 | 3
Not completed — Lost to Follow-up | 2 | 3
Period: Intervention
Arm/Group | Peer Coach Guided Online Learning Program | Self-administered Online Learning Program (Control)
Started | 47 | 49
Completed | 38 | 42
Not Completed | 9 | 7
Not completed — Physician Decision | 2 | 1
Not completed — Withdrawal by Subject | 5 | 6
Not completed — Lost to Follow-up | 2 | 0
Period: 1-Week Post-Intervention Data Collection
Arm/Group | Peer Coach Guided Online Learning Program | Self-administered Online Learning Program (Control)
Started | 38 | 42
Completed | 38 | 40
Not Completed | 0 | 2
Not completed — Lost to Follow-up | 0 | 2
Period: 3-Months Post-Intervention
Arm/Group | Peer Coach Guided Online Learning Program | Self-administered Online Learning Program (Control)
Started | 38 | 40
Completed | 38 | 38
Not Completed | 0 | 2
Not completed — Lost to Follow-up | 0 | 2

BASELINE CHARACTERISTICS:
Population: Subjects who were enrolled and randomized but did not complete baseline were excluded from analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | Peer Coach Guided Online Learning Program | Self-administered Online Learning Program (Control) | Total
Number analyzed (Participants) | 47 | 49 | 96
Age, Continuous [Mean (Standard Deviation); unit: Years] | 58.11 (7.22) | 57.18 (8.24) | 57.64 (7.73)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42 | 46 | 88
  Male | 5 | 3 | 8
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: White | 30 | 36 | 66
  Race/Ethnicity: Hispanic/Latinx | 5 | 4 | 9
  Race/Ethnicity: Black or African American | 7 | 5 | 12
  Race/Ethnicity: Asian/Pacific Islander | 2 | 1 | 3
  Race/Ethnicity: Native American or Alaskan Native | 2 | 0 | 2
  Race/Ethnicity: Other | 0 | 1 | 1
  Race/Ethnicity: Multiple Race/Ethnicity Selected | 1 | 2 | 3
Routine Assessment of Patient Index Data 3 (RAPID3) [Mean (Standard Deviation); unit: Units on a Scale] — RAPID3 is a questionnaire focusing on physical function, pain, and patient global assessment of disease activity. The score helps rheumatologists understand the impact of RA on daily life and can guide treatment decisions. A conversion table is used to simplify patient's weighed RAPID3 score. A score between 0 to 1.0 is defined as near remission (NR), 1.3 - 2 as low severity (LS), 2.3 - 4 as moderate severity (MS), and 4.3 - 10 as high severity (HS).
  Units on a Scale | 7.72 (6.62) | 7.14 (5.55) | 7.43 (6.07)
MOS Social Support Survey [Mean (Standard Deviation); unit: Units on a Scale] — Medical Outcomes Study (MOS) Social Support Survey consists of 19 questions that are averaged to compute a single score ranging from 1-5. The raw score is then transformed so that the final score ranges from minimum of 0 to maximum of 100 through the formula: 100 X [(observed score - minimum possible score)/(maximum possible score - minimum possible score)]. A higher score indicates more support. A score of 70 or higher indicates high support.
  Units on a Scale | 65.12 (23.69) | 63.93 (23.33) | 64.52 (23.39)
Patient Activation Measure (PAM-13) [Mean (Standard Deviation); unit: Units on a Scale] — Survey assesses patients' individual competencies for self-management. The mean score of the 13 items is calculated and transformed into a standardized activation score ranging from 0-100 based on a conversion table provided by the developers for data collected before 2014. The resulting 0-100 score is then used to categorize the individual into one of four levels of patient activation. The closer the score is to 100 the more activated a patient is.
  Units on a Scale | 43.26 (5.39) | 43.60 (6.40) | 43.43 (5.89)
PHQ-8 Patient Depression Questionnare [Mean (Standard Deviation); unit: Units on a Scale] — Depression measure for population based studies. Each question is on a scale from 0-3. Score is the sum of the 8 items. Lowest possible score is a 0 and the highest possible score is 24. A score of 10 or greater is considered major depression and 20 or more is severe major depression.
  Units on a Scale | 6.51 (4.87) | 7.29 (5.59) | 6.91 (5.23)
General Self-Efficacy Scale [Mean (Standard Deviation); unit: Units on a Scale] — A 10-item questionnaire designed to assess a person's optimistic self-belief in their ability to cope with a variety of difficult demands and stressful life events. The total score ranges from 10 to 40, with higher scores indicating higher self-efficacy. Scores above 30 indicate high generalized self-efficacy.
  Units on a Scale | 31 (5.20) | 30.42 (5.37) | 30.71 (5.27)
Medication Understanding and Use Self-Efficacy Scale (MUSE) [Mean (Standard Deviation); unit: Units on a Scale] — Survey measures self-efficacy of understanding and using prescription medication. Higher scores indicate a greater level of understanding and self-efficacy. Overall Muse scores range from 8-32. The average overall MUSE score is 30, so individuals scoring above 30 are categorized as having high medication understanding and use self-efficacy.
  Units on a Scale | 28.64 (5.39) | 27.88 (4.84) | 28.25 (5.11)

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Lipids Checked (Available Now Through National Laboratory Chain) or That Reported Having Their Lipids Checked by Their 1-week or 3-month Visit.
Description: Self-reported
Time Frame: 3 months post-intervention, approximately 20 weeks
Population: This analysis only includes individuals who had follow-up data.
Measure: Count of Participants; unit: Participants
Arm/Group | Peer Coach Guided Online Learning Program | Self-administered Online Learning Program (Control)
Number analyzed (Participants) | 38 | 38
Participants | 28 | 16
Statistical Analysis 1: Comparison: Peer Coach Guided Online Learning Program vs Self-administered Online Learning Program (Control); Test type: Superiority; p = 0.005, Chi-squared

2. Secondary Outcome: Change in General Self-Efficacy (GSF) Score From Baseline to the End of the Study Between Arms.
Description: The scale consists of 10 items and each item score ranges from 1 ("not at all true") to 4 ("exactly true"). Values 2 and 3 are assigned "barely true" and "moderately true", respectively. Scores are summed across the 10 items to give a total score, with a possible range of 10-40. Higher scores indicate greater confidence in generalized self-efficacy. Scores above 30 indicate high generalized self-efficacy, and scores 30 or below indicate low to moderate generalized self-efficacy.
  To find the change in GSF score from baseline to the end of the study between arms, the median of each participant's change in score was calculated.
Time Frame: Baseline and 3-months post-intervention, approximately 20 weeks
Population: This analysis only includes individuals who had follow-up data.
Measure: Median (Inter-Quartile Range); unit: Units on a Scale
Arm/Group | Peer Coach Guided Online Learning Program | Self-administered Online Learning Program (Control)
Number analyzed (Participants) | 38 | 38
Units on a Scale | 1 [-1 to 4] | 1 [0 to 5]
Statistical Analysis 1: Comparison: Peer Coach Guided Online Learning Program vs Self-administered Online Learning Program (Control); Test type: Superiority; p = 0.60, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Change in Patient Activation Measure (PAM) Score From Baseline to the End of the Study Between Arms.
Description: The scale consists of 13 items and each item score ranges from 0 ("not applicable") to 4 ("agree strongly"). Values 1, 2, and 3 are assigned "disagree strongly", "disagree", and "agree", respectively. Scores are summed across the 13 items to give a total score, with a range of 0-52. The mean score is then transformed into a standardized activation score ranging from 0-100, (the PAM score), based on a conversion table provided by the developer of the scale. Score ranges correspond to levels of activation, with higher levels indicating more activation: Level 1 - score of 47.0 or lower, Level 2 - score between 47.1 to 55.1, Level 3 - score between 55.2 to 72.4, Level 4 - score 72.5 or above.
  To find the change in PAM score from baseline to the end of the study between arms, the median of each participant's change in score was calculated.
Time Frame: Baseline and 3-months post-intervention, approximately 20 weeks
Population: Participants who did not complete 3-months survey were excluded from analysis.
Measure: Median (Inter-Quartile Range); unit: Units on a Scale
Arm/Group | Peer Coach Guided Online Learning Program | Self-administered Online Learning Program (Control)
Number analyzed (Participants) | 38 | 38
Units on a Scale | 1 [-2 to 4] | 1 [-1 to 6]
Statistical Analysis 1: Comparison: Peer Coach Guided Online Learning Program vs Self-administered Online Learning Program (Control); Test type: Superiority; p = 0.40, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Change in Routine Assessment of Patient Index Data (RAPID3) Score From Baseline to the End of the Study Between Arms.
Description: The scale consists of 12 score-able items. The scores from item 1 through 10, 11, and 12 are summed with a range of 0-30 and this is the RAPID3 cumulative score. A final conversion table is used to simplify the score. A score between 0-1.0 is defined as near remission (NR); 1.3-2.0 is low severity (LS); 2.3-4.0 is moderate severity (MS); and 4.3-10.0 is high severity (HS).
  To find the change in RAPID3 score from baseline to the end of the study between arms, the median of each participant's change in score was calculated.
Time Frame: Baseline and 3-months post-intervention, approximately 20 weeks
Population: This analysis only includes individuals who had follow-up data.
Measure: Median (Inter-Quartile Range); unit: Units on a Scale
Arm/Group | Peer Coach Guided Online Learning Program | Self-administered Online Learning Program (Control)
Number analyzed (Participants) | 38 | 38
Units on a Scale | 0.00 [-0.53 to 0.83] | -0.10 [-0.47 to 0.50]
Statistical Analysis 1: Comparison: Peer Coach Guided Online Learning Program vs Self-administered Online Learning Program (Control); Test type: Superiority; p = 0.60, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Change in Patient Health Questionnaire - 8 (PHQ-8) Score From Baseline to the End of the Study Between Arms
Description: The scale consists of 8 items, and each item score ranges from 0 ("not at all") to 3 ("nearly every day"). Scores are summed across the 8 items. The lowest possible score is 0 and the highest possible is 24. A score of 10 or greater is considered major depression and 20 or more is severe major depression.
  To find the change in PHQ-8 score from baseline to the end of the study between arms, the median of each participant's change in score was calculated.
Time Frame: Baseline and 3-months post-intervention, approximately 20 weeks
Population: This analysis only includes individuals who had follow-up data.
Measure: Median (Inter-Quartile Range); unit: Units on a Scale
Arm/Group | Peer Coach Guided Online Learning Program | Self-administered Online Learning Program (Control)
Number analyzed (Participants) | 38 | 38
Units on a Scale | -1 [-3 to 1] | 0 [-3 to 1]
Statistical Analysis 1: Comparison: Peer Coach Guided Online Learning Program vs Self-administered Online Learning Program (Control); Test type: Superiority; p = 0.50, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: Change in MOS Social Support Survey Score From Baseline to the End of the Study Between Arms.
Description: The survey consists of 4 separate social support sub-scales and an overall functional social support index for a total of 19 items. To obtain an overall support index score, the average is calculated for both the first 18 items in the scale and the last item in the scale from a range of 1-5. Scale scores are transformed to a 0-100 scale using a formula. A higher score indicates more support. The average score for the overall support index is 70, so individuals scoring above 70 are categorized as having high support and individuals scoring 70 or lower are categorized as having low to moderate support.
  To find the change in social support survey score from baseline to the end of the study between arms, the median of each participant's change in score was calculated.
Time Frame: Baseline and 3-months post-intervention, approximately 20 weeks
Population: This analysis only includes individuals who had follow-up data.
Measure: Median (Inter-Quartile Range); unit: Units on a Scale
Arm/Group | Peer Coach Guided Online Learning Program | Self-administered Online Learning Program (Control)
Number analyzed (Participants) | 38 | 38
Units on a Scale | 1 [-4 to 9] | 2 [-4 to 9]
Statistical Analysis 1: Comparison: Peer Coach Guided Online Learning Program vs Self-administered Online Learning Program (Control); Test type: Superiority; p = 0.90, Wilcoxon (Mann-Whitney)

7. Secondary Outcome: Change in Medication Understanding and Use Self-Efficacy Scale (MUSE) Score From Baseline to the End of the Study Between Arms.
Description: The scale consists of 8 items. Possible scores for overall MUSE range from 8-32. A higher overall MUSE score indicates a higher level of self-efficacy in understanding and using prescription medications. The average overall MUSE score is 30, so individuals scoring above 30 are categorized as having high medication understanding and use self-efficacy and individuals scoring 30 or lower are categorized as having low to moderate medication understanding and use self-efficacy.
  To find the change in MUSE scale scoring from baseline to the end of the study between arms, the median of each participant's change in score was calculated.
Time Frame: Baseline and 3-months post-intervention, approximately 20 weeks
Population: This analysis only includes individuals who had follow-up data.
Measure: Median (Inter-Quartile Range); unit: Units on a Scale
Arm/Group | Peer Coach Guided Online Learning Program | Self-administered Online Learning Program (Control)
Number analyzed (Participants) | 38 | 38
Units on a Scale | 0 [-1 to 1] | 0 [0 to 2]
Statistical Analysis 1: Comparison: Peer Coach Guided Online Learning Program vs Self-administered Online Learning Program (Control); Test type: Superiority; p = 0.20, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: From enrollment up to approximately 17 weeks
Arm/Group | Peer Coach Guided Online Learning Program | Self-administered Online Learning Program (Control)
All-Cause Mortality (participants affected / at risk) | 0/49 | 0/52
Serious Adverse Events (participants affected / at risk) | 0/49 | 0/52
Other Adverse Events (participants affected / at risk) | 1/49 | 1/52
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Peer Coach Guided Online Learning Program (N=49) | Self-administered Online Learning Program (Control) (N=52)
Inappropriate Behavior Towards Coach (Social circumstances) | 1 (1) | 0 (0) — Participant had to be removed for aggressive behavior toward peer coach
Alarmingly High PHQ-8 Score (Social circumstances) | 0 (0) | 1 (1) — Participant's PHQ fell into severely depressed category that physician though it best to remove them from the program

LIMITATIONS AND CAVEATS:
Because of our sample size, there is not a large enough power to make calculations that are statistically significant. Recruitment originally proved difficult because of the eligibility criteria requiring participants to not have had or discussed a cholesterol test due to participant's ambivalence on their certainty of having had one. This criterion was later removed two years into the study to ease recruitment. Intervention being anchored around physician's appointment also limited eligibility.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-02-06): https://cdn.clinicaltrials.gov/large-docs/97/NCT04488497/Prot_SAP_000.pdf